CLINICAL TRIAL: NCT06283888
Title: Safety and Efficacy of CYP2C19 Genotype-Guided P2Y12 Receptor Inhibitor Selection Versus Conventional Antiplatelet Therapy After Complex Percutaneous Coronary Intervention: The PRECISE-PCI Randomized Clinical Trial
Brief Title: CYP2C19 Genotype-Guided P2Y12 Receptor Inhibitor Selection After Complex Percutaneous Coronary Intervention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Cai De Jin, MD, MD, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRECISE-PCI
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: ACS - Acute Coronary Syndrome; CYP2C19 Polymorphism
Keywords: CYP2C19 Genotype; P2Y12 Receptor Inhibitor; Complex PCI
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYP2C19 Genotype Guided DAPT (Experimental): Patients with CYP2C19 *2 or *3 carrier will be received ticagrelor 60mg or 45mg bid (if <50 kg, ≥75 years) + aspirin 100 mg Patients with CYP2C19 *2 or *3 non-carrier will be received clopidogrel 75mg qd + aspirin 100 mg qd
  At post-PCI 3 months, monotherapy P2Y12 inhibitor (ticagrelor or clopidogrel) will be treated for a further 9 months.
  Interventions: Drug: CYP2C19 Genotype Guided DAPT
- Conventional DAPT (Experimental): Patients will be conventionally received ticagrelor 90mg bid or clopidogrel 75mg qd + aspirin 100 mg qd
  At post-PCI 3 months, monotherapy P2Y12 inhibitor (ticagrelor or clopidogrel) will be treated for a further 9 months.
  Interventions: Drug: Conventional DAPT

INTERVENTIONS:
Drug: CYP2C19 Genotype Guided DAPT — Patients with *2 or *3 carrier will be received ticagrelor 60mg or 45mg bid (if <50 kg, ≥75 years) + aspirin 100 mg qd; Patients with *2 or *3 non-carrier will be received clopidogrel 75mg qd + aspirin 100 mg qd
  Other Names: Guided DAPT
  Arms: CYP2C19 Genotype Guided DAPT
Drug: Conventional DAPT — Patients will be conventionally received ticagrelor 90mg bid or clopidogrel 75mg qd + aspirin 100 mg qd
  Other Names: Unguided DAPT
  Arms: Conventional DAPT

SUMMARY:
In Ease Asia clinical trials, P2Y12 inhibitor (ticagrelor or clopidogrel) monotherapy after 3-month dual antiplatelet therapy (DAPT) resulted in a lower incidence of clinically significant bleeding, without increasing risk of major adverse cardiac and cerebrovascular events, even if acute coronary syndrome (ACS) following complex percutaneous coronary intervention (PCI) when compared with standard DAPT. Although better understood "East Asian Paradox", finding the right CYP2C19 genotype-guided P2Y12 inhibitor selection to balance maintaining ischaemic prevention and less bleeding remains a topic in real-world clinical practice.

DETAILED DESCRIPTION:
In the PRECISE-PCI (CYP2C19 Genotype-Guided P2Y12 RECeptor Inhibitor SElection After Complex PCI) trial, the investigators aim to evaluate the safety and efficacy of CYP2C19 genotype-guided P2Y12 receptor inhibitor selection, as compared with conventional therapy in Chinese with ACS undergoing complex PCI All eligible ACS patients will be received DAPT (ticagrelor 180 mg or clopidogrel 300/600 mg plus aspirin 300 mg loading) before PCI. Subsequently to be randomly assigned into the genotype-guided group (CPY2C19 *2 or *3 carrier: ticagrelor 60 mg bid, or 45mg bid if <50 kg, ≥75 years; CPY2C19 *2 or *3 non-carrier: clopidogrel 75 mg qd in combination with aspirin 100 mg qd) and conventional group (ticagrelor 90 mg bid or clopidogrel 75 mg qd in combination with aspirin 100 mg qd). At post-PCI 3 months, both groups will be treated with mono-ticagrelor/clopidogrel without aspirin therapy for a further 9 months.

The primary endpoint is focusing on the net adverse clinical events (NACEs, a composite of cardiac death, non-fatal myocardial infarction, target vessel/lesion revascularization, stroke, or BARC-defined clinically significant bleeding type 2, 3, or 5) during 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Criteria:

   * Patients aged between 18-80 years old.
   * Patients with ACS (UA/NSTEMI/STEMI) undergoing PCI.
   * Patients will be treated with DAPT (P2Y12 inhibitors+aspirin) for at least 3 months.
   * Patients are willing to provide a DNA sample (via blood draw) for CYP2C19 genotyping.
   * Patients provide written informed consent before enrollment.
2. Angiographic Criteria (meet at least 1 of the following characteristics):

   * Thrombotic target lesion.
   * Calcified target lesion requiring rotational atherectomy or intravascular lithotripsy
   * Multivessel (≥2 vessels) disease will be treated.
   * Multi-target lesions (≥3 lesions) will be treated.
   * Multi-stent (≥3 stents) will be implanted.
   * Total stent length≥60 mm.
   * Bifurcation lesion requiring at least 2 stents.
   * PCI for left main.
   * PCI for chronic total occlusion.
   * PCI for bypass graft.

Exclusion Criteria:

* Patient with known CYP2C19 genotype before randomization.
* Anticipated discontinuation of clopidogrel or ticagrelor within the 12-month follow-up period.
* Planned surgery within 90 days.
* Requiring oral anticoagulation therapy (eg, atrial fibrillation, deep vein thrombosis, pulmonary thromboembolism)
* Intracranial/gastrointestinal/urogenital bleeding within 6 months.
* Active bleeding or bleeding diathesis, thrombocytopenia (platelet <100,000/mL) or hemoglobin <10 g/dL
* Hepatic dysfunction (serum liver enzyme>3 times the normal limit)
* Renal failure (eGFR <15 ml/min/1.73m2 or requiring dialysis)
* Concomitant therapy with a strong CYP3A4 inhibitor or inducer
* Life expectancy < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
NACE (net adverse clinical event) | At 12 months
  The incidence of NACE (composite of cardiac death, non-fatal myocardial infarction, target vessel/lesion revascularization, stroke, or clinically significant bleeding according to BARC criteria).

SECONDARY OUTCOMES:
Incidence of clinically significant bleeding | At 12 months
  The Bleeding Academic Research Consortium (BARC)-defined clinically significant bleeding (type 2, 3, or 5 bleeding) as follows:
  Type 2: Any overt, actionable sign of hemorrhage, requiring nonsurgical, medical intervention by a healthcare professional; Leading to hospitalization or increased level of care; Prompting evaluation.
  Type 3: Clinical, laboratory, and/or imaging evidence of bleeding with specific healthcare provider responses.
  Type 3a: Overt bleeding plus hemoglobin drop of 3 to 5 g/dL; Any transfusion with overt bleeding.
  Type 3b: Overt bleeding plus hemoglobin drop ≥5 g/dL; Cardiac tamponade; Bleeding requiring surgical intervention for control; Bleeding requiring intravenous vasoactive agents.
  Type 3c: Intracranial hemorrhage; Subcategories confirmed by autopsy or imaging or lumbar puncture; Intraocular bleed compromising vision.
  Type 5: Fatal bleeding is bleeding that directly causes death with no other explainable cause.
Incidence of MACCE | 12 months
  The incidence of major adverse cardiac and cerebrovascular event (MACCE), is composite of cardiac death, non-fatal myocardial infarction, target vessel/lesion revascularization, or stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Cai De Jin, Principal Investigator — Zunyi Medical College
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

REFERENCES:
- [Background] Pereira NL, Farkouh ME, So D, Lennon R, Geller N, Mathew V, Bell M, Bae JH, Jeong MH, Chavez I, Gordon P, Abbott JD, Cagin C, Baudhuin L, Fu YP, Goodman SG, Hasan A, Iturriaga E, Lerman A, Sidhu M, Tanguay JF, Wang L, Weinshilboum R, Welsh R, Rosenberg Y, Bailey K, Rihal C. Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy on Ischemic Outcomes After Percutaneous Coronary Intervention: The TAILOR-PCI Randomized Clinical Trial. JAMA. 2020 Aug 25;324(8):761-771. doi: 10.1001/jama.2020.12443. PMID 32840598
- [Background] Kim BK, Hong SJ, Cho YH, Yun KH, Kim YH, Suh Y, Cho JY, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon H, Ahn CM, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; TICO Investigators. Effect of Ticagrelor Monotherapy vs Ticagrelor With Aspirin on Major Bleeding and Cardiovascular Events in Patients With Acute Coronary Syndrome: The TICO Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2407-2416. doi: 10.1001/jama.2020.7580. PMID 32543684
- [Background] Hahn JY, Song YB, Oh JH, Chun WJ, Park YH, Jang WJ, Im ES, Jeong JO, Cho BR, Oh SK, Yun KH, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Lee WS, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC; SMART-CHOICE Investigators. Effect of P2Y12 Inhibitor Monotherapy vs Dual Antiplatelet Therapy on Cardiovascular Events in Patients Undergoing Percutaneous Coronary Intervention: The SMART-CHOICE Randomized Clinical Trial. JAMA. 2019 Jun 25;321(24):2428-2437. doi: 10.1001/jama.2019.8146. PMID 31237645
- [Background] Jin C, Kim MH, Guo LZ, Jin E, Shin ES, Ann SH, Cho YR, Park JS, Kim SJ, Lee MS. Pharmacodynamic study of prasugrel or clopidogrel in non-ST-elevation acute coronary syndrome with CYP2C19 genetic variants undergoing percutaneous coronary intervention (PRAISE-GENE trial). Int J Cardiol. 2020 Apr 15;305:11-17. doi: 10.1016/j.ijcard.2020.01.058. Epub 2020 Jan 25. PMID 32029306
- [Background] Jin CD, Kim MH, Song K, Jin X, Lee KM, Park JS, Cho YR, Yun SC, Lee MS. Pharmacodynamics and Outcomes of a De-Escalation Strategy with Half-Dose Prasugrel or Ticagrelor in East Asians Patients with Acute Coronary Syndrome: Results from HOPE-TAILOR Trial. J Clin Med. 2021 Jun 18;10(12):2699. doi: 10.3390/jcm10122699. PMID 34207339